CLINICAL TRIAL: NCT04206111
Title: Evaluation of Gastric Insufflation Measured by Ultrasound of the Antral Surface During Optiflow Preoxygenation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Other Study IDs: Optisafe
Record Dates: First submitted 2019-12-15; First posted 2019-12-20 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Gastric Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preoxygenation
  Interventions: Procedure: Preoxygenation

INTERVENTIONS:
Procedure: Preoxygenation — preoxygenation with high flow nasal cannula at 40l/min for 5min

SUMMARY:
Check in gastric ultrasound for lack of stomach insufflation during preoxygenation with high-flow nasal cannulas

ELIGIBILITY:
Inclusion Criteria:

* Adults Volunteers

Exclusion Criteria:

* History of gastric surgery
* Facial or oropharyngeal abnormality

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
no gastric insufflation | From date of randomization until the date of first documented progression, whichever came first, assessed up to 6 months
  Number of Participants with no gastric insufflation

CONTACTS AND LOCATIONS:
Locations (1):
- Javillier, Liège, Belgium